CLINICAL TRIAL: NCT01231997
Title: Clinical Study to Investigate the Safety and Pharmacokinetics of Udenafil Tablet in Renal Impaired Male Patients
Acronym: DA8159_RI_I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Clinical Development Team1, Dong-A Pharmaceutical Co., Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0431
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Renal Insufficiency; Kidney Diseases; Urologic Diseases
Keywords: Udenafil; DA-8159; renal impairment; healthy volunteers
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Urologic Diseases | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental)
  Interventions: Drug: Udenafil
- Patients with mild renal impairment (Experimental)
  Interventions: Drug: Udenafil
- Patients with moderate renal impairment (Experimental)
  Interventions: Drug: Udenafil
- Patients with severe renal impairment (Experimental)
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — 100mg Single Oral Dose of

SUMMARY:
This study is designed to assess the effect of renal impairment on the pharmacokinetics, safety and tolerability of udenafil in subjects with renal impairment compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 19 to 64 years at screening.
* Subjects with body weight ≥ 55 kg and within ±30% of the ideal body weight : Ideal body weight = (height [cm] - 100)x0.9.
* Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

* Subjects with the test results of QTc > 430 ms or non-sinus cardiac rhythm by ECG analysis.
* Subjects with hypotension or hypertension.
* Subjects who have drunken habitually (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the study period from 2 days prior to the first administration of investigational product and during this study.
* Subjects deemed ineligible by investigator based on other reasons, including abnormal laboratory values or diseases.

Ages: 19 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax) | up to 48 hours

SECONDARY OUTCOMES:
Safety | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr